CLINICAL TRIAL: NCT05996783
Title: Cervical Cancer Screening Based on First-void Urine Self-sampling to Reach un(Der)-Screened Women: ScreenUrSelf Trial
Acronym: ScreenUrSelf
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Antwerp University Hospital (UZA) (Unknown); Centre for Cancer Detection (CvKO) (Unknown); Sciensano (Other Government)
Responsible Party: Principal Investigator, Pierre Van Damme, Principal Investigator, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B3002023000026
Record Dates: First submitted 2023-08-02; First posted 2023-08-18 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Cervix Cancer; Cervical Intraepithelial Neoplasia; Human Papilloma Virus; HPV-Related Cervical Carcinoma
Keywords: Biomarker; First-void urine; Vaginal sample; Screening; Triage; Self-sampling; Prevention
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Control - no intervention (No Intervention): This control group will receive no intervention. Cervical cancer screening (having a Pap smear taken by a clinician for cytology-based screening) is completely opportunistic, i.e. based on the initiative of the participant or their clinician.
  No reminder letter will be sent.
- Control - (recall) invitation letter (No Intervention): This control group will receive the standard (recall) invitation letter send out by the Centre for Cancer Detection (CvKO). In this invitation letter, participants are encouraged to make an appointment with their clinician to have a Pap smear taken (for cytology-based screening).
  A reminder letter will be sent after 5-6 months.
- Opt-out first-void urine (Experimental): Women will receive a first-void urine self-sampling study package at home.
  The study package will include an invitation letter/informed consent form, information brochure, first-void urine self-sampling device, safety bag with absorbent paper, pre-stamped return envelope, and instructions explaining how to collect the sample and send it to the lab.
  A reminder letter will be sent after 5-6 months.
  Interventions: Device: Colli-Pee Small Volumes
- Opt-in first-void urine (Experimental): Women will receive a letter at home with instructions how to order (via phone, e-mail, or webform) a first-void urine self-sampling study package.
  The study package will include an invitation letter/informed consent form, information brochure, first-void urine self-sampling device, safety bag with absorbent paper, pre-stamped return envelope, and instructions explaining how to collect the sample and send it to the lab.
  A reminder letter will be sent after 5-6 months.
  Interventions: Device: Colli-Pee Small Volumes
- Opt-out vaginal self-sample (Experimental): Women will receive a vaginal self-sampling study package at home.
  The study package will include an invitation letter/informed consent form, information brochure, vaginal self-sampling device, safety bag with absorbent paper, pre-stamped return envelope, and instructions explaining how to collect the sample and send it to the lab.
  A reminder letter will be sent after 5-6 months.
  Interventions: Device: Evalyn Brush
- Opt-in vaginal self-sample (Experimental): Women will receive a letter at home with instructions how to order (via phone, e-mail, or webform) a vaginal self-sampling study package.
  The study package will include an invitation letter/informed consent form, information brochure, vaginal self-sampling device, safety bag with absorbent paper, pre-stamped return envelope, and instructions explaining how to collect the sample and send it to the lab.
  A reminder letter will be sent after 5-6 months.
  Interventions: Device: Evalyn Brush

INTERVENTIONS:
Device: Colli-Pee Small Volumes — Women will self-collect a first-void urine sample at home upon receipt of the study package using the Colli-Pee Small Volumes (10 mL) device (Novosanis, Belgium). The collector tube is prefilled with a preservative (UCM, Novosanis, Belgium). Women will send the collector vial containing first-void urine along with the informed consent form to the laboratory at University of Antwerp using the prestamped envelope.
  Arms: Opt-in first-void urine; Opt-out first-void urine
Device: Evalyn Brush — Women will self-collect a vaginal sample at home upon receipt of the study package using the Evalyn Brush device (Rovers Medical Devices, The Netherlands). Women will send the used brush along with the informed consent form to the laboratory at University of Antwerp using the prestamped envelope.
  Arms: Opt-in vaginal self-sample; Opt-out vaginal self-sample

SUMMARY:
The goal of the ScreenUrSelf trial is to increase cervical cancer screening attendance and compliance to follow-up by offering a first-void urine self-sampling alternative to women who are currently not participating in the organized cervical cancer screening program (defined in this project as un(der)-screened women), either on the woman or her physician's personal initiative, or by responding on the invitation letter.

DETAILED DESCRIPTION:
Patient: In this population-based study we target real un(der)-screened women, i.e., women (31-64y) eligible for the Flemish population-based cervical cancer screening program without any cytology/histology/pathological result retrieved from the Belgian Cancer Registry (BCR) for at least the last six years (i.e., two screening rounds). Women who opted out of the screening program, who are pregnant (self-reported), underwent total hysterectomy, have (had) cervical or uterine cancer, or are included in other Centre for Cancer Detection (CvKO) pilot projects are not eligible.

Intervention: The proposed randomized controlled trial (RCT) will be embedded in the Flemish organized cervical cancer screening program, which is coordinated by CvKO under governance of the Flemish government. The goal is to reach women who are eligible but do not participate in cervical cancer screening, by offering two self-sampling methods (first-void urine and vaginal) in an opt-in and -out strategy (total of four interventions) to collect samples for primary high-risk (hr) Human Papillomavirus (HPV) testing, and if positive, reflex 1) cytology on a Pap smear (standard of care) and 2) methylation marker triage (index test).

Comparison: The two control arms include 1) no intervention; and 2) sending (recall) invitation letters to women, inviting them to make an appointment for a Pap smear (i.e., current practise within the organized cervical cancer screening program in Flanders).

Primary outcome: The primary outcome is the actual response rate, i.e., proportions of women that participate in each intervention and in the control arms at 12 months after initiation of the intervention (the intervention being one of six study arms). Response in this project is defined as having a preventive cervical screen exam, either by a self-sample or by a physician-taken Pap smear, at 12 months after initiation of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for cervical cancer screening within the organized Population-based Screening Program in Flanders:

  * Female
  * Residing in Flanders, Belgium
  * Not actively opted out of the organized cervical cancer screening program
  * No history of total hysterectomy (data available since 2002)
  * No (former) diagnosis of cervical or uterine cancer (data available as of 2008)
  * Not included in other CvKO pilot projects
* No cervical result registered in the cytohistopathological register of BCR and no information in the administrative data from health insurance companies (IMA) on PAP smears taken for at least the last 6 years (i.e., two screening rounds)
* 31-64 years old (birth year 1959-1992)

Exclusion Criteria:

* Being pregnant or 6 weeks postpartum (self-reported after receiving the study letter/package)
* Participation during menstruation or within the 3 following days is a contraindication
* Not able to understand the study materials and participation form (informed consent form)

Ages: 31 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48000 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Response rate | 10 months (until 31/03/2024)
  Proportions of women that participate in each intervention (measured by PP* and ITT*) and in the control arms (measured by Pap smears taken) within 10 months after the intervention.
  *PP: participation in intervention arm measured by self-sample analyses only
  **ITT: participation in intervention arm measured by self-sample analyses or Pap smears taken

SECONDARY OUTCOMES:
Compliance | 19 months (until 31/12/2024)
  1. Compliance to a hrHPV positive result on a self-sample measured by standard of care follow-up, i.e., a Pap smear taken by a clinician.
  2. Compliance to an abnormal Pap smear measured by standard of care follow-up.
Preference | Through study completion, an average of 1 year
  Preference and attitudes of women between intervention arms (measured via a questionnaire)
Age-related differences in response rate | 10 months (until 31/03/2024)
  Age-related differences in response rates within and between different study arms
  Response rates: Proportions of women that participate in each intervention (measured by PP* and ITT*) and in the control arms (measured by Pap smears taken) within 10 months after the intervention.
  *PP: participation in intervention arm measured by self-sample analyses only
  **ITT: participation in intervention arm measured by self-sample analyses or Pap smears taken
Socio-economic status-related differences differences in response rate | 10 months (until 31/03/2024)
  Socio-economic status-related differences in response rates within and between different study arms
  Response rates: Proportions of women that participate in each intervention (measured by PP* and ITT*) and in the control arms (measured by Pap smears taken) within 10 months after the intervention.
  *PP: participation in intervention arm measured by self-sample analyses only
  **ITT: participation in intervention arm measured by self-sample analyses or Pap smears taken
Clinical accuracy of HPV assay | Through study completion, an average of 1 year
  Test-positivity, positive predictive value, referral rate to colposcopy, and detection rate of CIN2+ of a hrHPV positive result on a self-sample in un(der)-screened women; absolute measures in each arm and ratios of measures between arms.
  Test-positivity, positive predictive value, referral rate to colposcopy, and detection rate of CIN2+ will be combined to report clinical accuracy.
Clinical accuracy of methylation assay | Through study completion, an average of 1 year
  Test-positivity, positive predictive value, referral rate to colposcopy, and detection rate CIN2+ of a methylation-based reflex test (index test) to triage hrHPV positive self-sample in un(der)screened women, compared to reflex cytology on a Pap smear (comparator test); absolute measures in each arm and ratios of measures between arms.
  Test-positivity, positive predictive value, referral rate to colposcopy, and detection rate of CIN2+ will be combined to report clinical accuracy.
Cost-effectiveness | Through study completion, an average of 1 year
  1. Differences in time needed per women to obtain a test result between study arms
  2. Differences in costs per women between the different study arms
  3. Differences in total cost between the different study arms
  The above differences in time and costs will be combined to report cost-effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Van Damme, MD, PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Universiteit Antwerpen, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No